CLINICAL TRIAL: NCT02533804
Title: A Community Epidemiology Study Evaluating the Factors Influencing Overall Health and Wellness
Brief Title: The Lake Nona Life Project
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Collaborators: Lake Nona Institute (Unknown); DataStat, Inc. (Unknown); Mytrus, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1166275
Record Dates: First submitted 2015-06-01; First posted 2015-08-27 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Health Behavior; Quality of Life; Aging
Keywords: health; wellness; life expectancy; quality of life; performance; religion; skin; cardiovascular; joints; bone; respiration; pain; nervous system diseases; oral health; behavior; child; depression; mood; panic; sleep; stress; nutrition; exercise; life change events; personality; employment; social networking; time management; residence characteristics
MeSH Terms: conditions — Health Behavior; Respiratory Aspiration; Pain; Nervous System Diseases; Behavior; Depression; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Lake Nona Life Project aims to examine the health and wellness of participants over the course of multiple years, focusing on the links between health and wellness, longevity, quality of life, and human performance.

DETAILED DESCRIPTION:
The Lake Nona Life Project is a community health and wellness research project of the Lake Nona Institute (LNI), carried out by the Lake Nona Medical City Residents and Partners (the Researchers), and sponsored by Florida Hospital. The project is designed to study patterns, predictors and strategies for improving human health and wellness. Data will be obtained over many years using surveys/interviews, medical tests, and health information from 3rd parties (i.e., health care claims data) obtained with participant permission.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Live and/or work in the Lake Nona Community (proper)
* Able to provide informed consent
* Able to speak and read English

Exclusion Criteria:

* Unable to speak or communicate in English
* Living outside of the LNLP study map
* Cognitive impairment that would not allow survey completion
* Unable to speak and read English

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults ages 18 and older living and/or working in the Lake Nona Community (proper) of Orlando, Florida.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-12-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life over 10 Years | 20 years
  Participants will self report on an Investigator created questionnaire regarding life satisfaction, stress and life events. Responses will be provided on a five point Likert Scale.

SECONDARY OUTCOMES:
Demographics | 20 years
  Participants will self report demographic information consisting of questions related to age, gender and race.
Medical History | 20 years
  Participants will self report medical history and chronic conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Robinson, Principal Investigator — Center for CREATION Health Research
Locations (1):
- Lake Nona Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Institute for Health Metrics and Evaluation. 2013. Financing Global Health 2012: The End of the Golden Age? Seattle, WA: IHME http://www.healthmetricsandevaluation.org/publications/policy-report/financing-global-health-2012-end-golden-age
- [Background] World Health Organization. (2012). World Health Statistics 2012. Geneva, Switzerland: World Health Organization http://www.who.int/gho/publications/world_health_statistics/EN_WHS2012_TOC.pdf?ua=1
- [Background] United Nations, Department of Economic and Social Affairs, Population Division. (2011). World population prospects, the 2010 revision. http://esa.un.org/unpd/wpp/Documentation/WPP%202010%20publications.htm
- [Background] Organization for Exonomic Co-operation and Development. (2012). OECD Health Data 2012: U. S. Health Care System from an International Perspective [PDF document]. Retrieved from http://www.oecd.org/health/HealthSpendingInUSA_HealthData2012.pdf
- [Background] US Central Intelligence Agency. (2014). The World Factbook, Country Comparison: Life Expectancy at Birth. Retrieved from https://www.cia.gov/library/publications/the-world-factbook/rankorder/2102rank.html
- [Background] Murphy SL, Xu J, Kochanek KD. Deaths: final data for 2010. Natl Vital Stat Rep. 2013 May 8;61(4):1-117. PMID 24979972
- [Background] Rand Health. (2000). Projection of chronic illness prevalence and cost inflation. Santa Monica, CA: Wu, S., Y., Green, A.
- [Background] Kung HC, Hoyert DL, Xu J, Murphy SL. Deaths: final data for 2005. Natl Vital Stat Rep. 2008 Apr 24;56(10):1-120. PMID 18512336
- [Background] National Center for Chronic Disease Prevention and Health Promotion. (2012). Chronic Diseases and Health Promotion. Retrieved from http://www.cdc.gov/chronicdisease/overview/index.htm
- [Background] Adams PF, Kirzinger WK, Martinez ME. Summary health statistics for the u.s. Population: national health interview survey, 2011. Vital Health Stat 10. 2012 Dec;(255):1-110. PMID 25116371
- [Background] National Heart, Lung, and Blood Institute, Boston University. (2014). The Framingham Heart Study Bibliography. Retrieved from http://www.framinghamheartstudy.org/fhs-bibliography/index.php
- [Background] Cranor CW, Bunting BA, Christensen DB. The Asheville Project: long-term clinical and economic outcomes of a community pharmacy diabetes care program. J Am Pharm Assoc (Wash). 2003 Mar-Apr;43(2):173-84. doi: 10.1331/108658003321480713. PMID 12688435
- [Background] Bunting BA, Cranor CW. The Asheville Project: long-term clinical, humanistic, and economic outcomes of a community-based medication therapy management program for asthma. J Am Pharm Assoc (2003). 2006 Mar-Apr;46(2):133-47. doi: 10.1331/154434506776180658. PMID 16602223
- [Background] Bunting BA, Smith BH, Sutherland SE. The Asheville Project: clinical and economic outcomes of a community-based long-term medication therapy management program for hypertension and dyslipidemia. J Am Pharm Assoc (2003). 2008 Jan-Feb;48(1):23-31. doi: 10.1331/JAPhA.2008.07140. PMID 18192127
- [Background] Luepker RV, Murray DM, Jacobs DR Jr, Mittelmark MB, Bracht N, Carlaw R, Crow R, Elmer P, Finnegan J, Folsom AR, et al. Community education for cardiovascular disease prevention: risk factor changes in the Minnesota Heart Health Program. Am J Public Health. 1994 Sep;84(9):1383-93. doi: 10.2105/ajph.84.9.1383. PMID 8092360
- [Background] Belloc NB, Breslow L. Relationship of physical health status and health practices. Prev Med. 1972 Aug;1(3):409-21. doi: 10.1016/0091-7435(72)90014-x. No abstract available. PMID 5085007
- [Background] GORDON T. Mortality experience among the Japanese in the United States, Hawaii, and Japan. Public Health Rep (1896). 1957 Jun;72(6):543-53. No abstract available. PMID 13432134
- [Background] Yano K, Reed DM, McGee DL. Ten-year incidence of coronary heart disease in the Honolulu Heart Program. Relationship to biologic and lifestyle characteristics. Am J Epidemiol. 1984 May;119(5):653-66. doi: 10.1093/oxfordjournals.aje.a113787. PMID 6720665
- See also: General Information/Registration — http://www.liveworkparticipate.com